CLINICAL TRIAL: NCT01663610
Title: Online Course for Adults With ADHD or Subclinical ADHD Teaching How to Use a Smartphone as a Support in Their Everyday Life
Brief Title: Online Course Teachning Adults With ADHD How to Use a Smartphone
Acronym: VardagsSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012334314
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VardagsSMART (Experimental): VardagsSMART Internet-based course with therapist support during 6 weeks
  Interventions: Behavioral: VardagsSMART
- Wait List Control (CONT) (No Intervention): Weekly registrations only. After 6 weeks the Internet-based course without therapist support well be offered (SelfSMART)

INTERVENTIONS:
Behavioral: VardagsSMART — VardagsSMART Internet-based course with therapist support during 6 weeks
  Arms: VardagsSMART

SUMMARY:
This study is a randomized controlled trial (RCT) to evaluate the effect of an internet-based, guided self-help course for individuals who have recivied an ADHD diagnsis or struggle with organizing daily life and/or easily get distracted. The course (vardagsSMART) teach the participants how to use a Smartphone to better organize their everday life and will be compared to a wait list control group (CONT) that later will recieve the same course without guidance from a supervisor(selfSMART). It is hypothesized that VardagsSMART will be superior to CONT on ability to organize everyday life and ADHD-symptoms, and that vardagsSMART will be superior to selfSMART on adherence, understanding and perecived usefullness.

DETAILED DESCRIPTION:
Smartphones have a potential to improve the life of individuals who have major problems with structure and remembrance of everyday tasks. The automation by smartphones of these tasks away from caregivers to the individual is a process that is both time saving and positive for the individuals sense of autonomy.

There is too little research to date to say with clarity that smartphones is this tool for most of the patient group but many patients with ADHD report that a smartphone system for organisation and remembrance is a key that helps many live a more meaningful life.

The best way to teach these skills has not yet been proven. There is a clear advantage with teaching courses concerning IT in an online setting since hyperlinks and other texts can be easily forwarded and the course participants can easily use premade calendars and other tools. This research will try to determine if this type of online course is helpful for these patients.

VardagsSMART is an online course which will be compared to a waiting list controll group (CONT) which weekly records how they manage their ADHD symptoms.

The main purpose of this study is to examine whether the VardagsSMART course have a positive effect for the patient group. An untreated control group is used to ensure that the effects are not only due to spontaneous improvement. The control group will afterwards be offered the course without therapist support (SelfSMART), in order to make a preliminary evaluation of the importance of therapist support.

ELIGIBILITY:
Inclusion Criteria:

* have problems organizing daily activity measured by more then 17 points on the ASRS questionaire item 1-4 and 7-11-
* has acces to a smartphone (android or iphone) with internet acces.
* at least 18 years
* speaks, writes and read Swedish
* can not foresee any practical barriers to participation.

Exclusion Criteria:

* has a high alcohol or drug use assessed by the AUDIT / DUDIT and assessment interview.
* somatic or psychiatric problems that are directly contraindicated or seriously hamper the implementation of the treatment (eg, psychotic disorders).
* have severe depression, defined as MADRS-S over 30 or suicidal risk judged by more than 4 points on the MADRS-S question 9 or according to the structured telephone assessment.
* currently undergoing some form of treatment that focuses on reducing symptoms of ADHD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in symptoms of inattention and concentration | 6 weeks (Post) and 9 months (FU)
  Adult Self Report Scale (ASRS), the subscale measuring inattention and concentration (item 1-4 and 7-11)

SECONDARY OUTCOMES:
Change (from baseline) in ADHD symptoms | 6 weeks (Post) and 9 months (FU)
  Adult Self Report Scale (ASRS), Full Scale
Change (from baseline) in dialy life function | 6 weeks (Post) and 9 months (FU)
  Sheehan Disability Scale (SDS)
Change (from baseline) in Depression and Anxiety | 6 weeks (Post) and 9 months (FU)
  Hospital Anxiety and Depression Scale (HADS)
Change (from baseline) in perecived stress | 6 weeks (Post) and 9 months (FU)
  Perceived Stress Scale-4 (PSS-4)

OTHER OUTCOMES:
Treatment evaluation and usage | Post-treatment (6 weeks)
  Questions on treatment satisfaction, adherence, and precevied usefullness of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Ph.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienehten (Internet Psychiatry Unit), Psykiatri Sydväst, SLSO Stockholm, Sweden, Stockholm, Stockholm County, Sweden